CLINICAL TRIAL: NCT00795717
Title: Human Immunodeficiency Virus (HIV), Arterial Dysfunction, Lipids, Lovaza (HALO) Trial
Acronym: HALO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LVZ111888; 011293-GSK Contract Reference#
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Cardiovascular Disease; HIV Infection
Keywords: HIV; cardiovascular risk; atherogenic lipid profile; brachial artery reactivity; omega three fatty acids
MeSH Terms: conditions — Cardiovascular Diseases; HIV Infections | interventions — Omacor; Capsules; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lovaza (Active Comparator): Lovaza, dietary counseling
  Interventions: Drug: Lovaza
- Placebo (Placebo Comparator): Placebo, dietary counseling
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lovaza — Lovaza at a dose of 4g per day with each 1g capsule containing approximately 465 mg of eicosapentaenoic acid (EPA) and 375 docosahexaenoic acid (DHA) for 12 weeks.
  Other Names: Omacor (omega-3-acid ethyl esters) capsules
  Arms: Lovaza
Drug: Placebo — 2 capsules given twice daily
  Other Names: corn oil
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether fish oil supplementation with Lovaza, formally known as Omacor will result in a significant reduction in serum triglyceride (TG), an increase in high density lipoproteins(HDL), and an improvement of endothelial dysfunction.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled, cross-over, clinical trial to determine the effect of fish oil supplementation with Lovaza® on triglyceride levels in HIV-infected subjects on HAART with elevated serum triglycerides. The sample size is 40 subjects. The total duration of the study is 28 weeks, with 12-week treatment periods separated by a 4-week washout. This study will be conducted at the Clinical Research Center at Tufts Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected men and women at least 18 years of age
* On stable HAART for previous three months and without anticipated changes in their HAART regimen throughout the duration of the study
* Fasting triglycerides > 150 mg/dl and < 1,500 mg/dl
* Participants may be on lipid lowering therapy; if on lipid lowering therapy, therapy must be stable for 8 weeks and cannot be changes during the course of the study
* Participants may be on beta blockers (e.g., Atenolol, Metoprolol, Propranolol), Estrogens (e.g.,Estinyl;Estrace;Estraderm) and Thiazides (water pills), however therapy with these agents must be stable for 8 weeks before starting the study and cannot be altered while on the study unless deemed medically necessary by the participant's medical provider and approved by Dr. Wanke
* Female participants of reproductive age must not be pregnant (negative test) or lactating at screening and throughout the trial and agree to use 2 methods of barrier contraception for the course of the trial and 2 months after the trial unless they are surgically sterilized (tubal ligation or hysterectomy), or post-menopausal with no menses for > 1 year
* Ability to provide consent

Exclusion Criteria:

* Plasma HIV-1 RNA > 10,000
* Previous history of atherosclerotic disease or diabetes mellitus
* Change in HAART regimen over three months prior to study entry
* Change in lipid lowering therapy within 2 months
* On chronic anticoagulants such as heparin or coumadin
* On fish oil, omega 3 supplements, or Omacor currently or during the past month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine A Wanke, MD, Principal Investigator — Tufts University School of Medicine
Locations (1):
- Tufts University School of Medicine, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Paranandi A, Asztalos BF, Mangili A, Kuvin J, Gerrior J, Sheehan H, Skinner SC, Tang AM, Wanke CA. Short communication: effects of omega-3 fatty acids on triglycerides and high-density lipoprotein subprofiles in HIV-infected persons with hypertriglyceridemia. AIDS Res Hum Retroviruses. 2014 Aug;30(8):800-5. doi: 10.1089/AID.2014.0005. PMID 24988179

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phone contact n=109 Screening n=51 Eligible n=42 Screen failed n=9 Declined participation n=1 Randomized to treatment first n=20 Randomized to placebo first n=21
Groups:
- Lovaza Then Placebo: Lovaza, dietary counseling
  Lovaza : Lovaza at a dose of 4g per day with each 1g capsule containing approximately 465 mg of eicosapentaenoic acid (EPA) and 375 docosahexaenoic acid (DHA) for 12 weeks vs. placebo 2 capsules given twice daily.
- Placebo Then Lovaza: Placebo, dietary counseling
  Placebo : 2 capsules given twice daily vs. Lovaza at a dose of 4g per day with each 1g capsule containing approximately 465 mg of eicosapentaenoic acid (EPA) and 375 docosahexaenoic acid (DHA) for 12 weeks
Period: Phase I Followed by Wash Out x 4 Weeks
Arm/Group | Lovaza Then Placebo | Placebo Then Lovaza
Started | 20 (Randomized to treatment first) | 21 (Randomized to placebo first)
Completed | 18 | 19
Not Completed | 2 | 2
Not completed — alcohol treatment | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Phase II
Arm/Group | Lovaza Then Placebo | Placebo Then Lovaza
Started | 18 | 19
Completed | 18 | 18
Not Completed | 0 | 1
Not completed — too busy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lovaza Then Placebo: Lovaza, dietary counseling
  Lovaza : Lovaza at a dose of 4g per day with each 1g capsule containing approximately 465 mg of eicosapentaenoic acid (EPA) and 375 docosahexaenoic acid (DHA) for 12 weeks.
- Placebo Then Lovaza: Placebo or Corn oil pill, dietary counseling
  Corn oil pill : 2 capsules given twice daily for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Lovaza Then Placebo | Placebo Then Lovaza | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51.5 [46.5 to 55.0] | 55.0 [44.0 to 58.0] | 52.0 [45.0 to 58.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 17 | 18 | 35
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline Mean Serum Triglyceride Level at Study End
Description: Change in Baseline (time 0) Mean Serum Triglyceride levels after 12 weeks of treatment or placebo
Time Frame: Baseline and 12 weeks
Population: Randomized, cross over design
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Lovaza: Lovaza, dietary counseling
  Lovaza : Lovaza at a dose of 4g per day with each 1g capsule containing approximately 465 mg of eicosapentaenoic acid (EPA) and 375 docosahexaenoic acid (DHA) for 12 weeks.
- Placebo: Corn oil, dietary counseling
  Corn oil : 2 capsules given twice daily
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 39 | 39
mg/dl | -103.0 (92.2) | -23.4 (60.8)

2. Secondary Outcome: Serum HDL Level
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Placebo: Placebo, dietary counseling
  Placebo : 2 capsules given twice daily
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 39 | 39
mg/dl | 39 (12) | 36 (10)

3. Secondary Outcome: Brachial Artery Reactivity
Description: To demonstrate the impact of omega-three fatty acid intake on BART (Brachial Artery Reactivity Test) at 12 weeks.
  Brachial artery ultrasound measurements Brachial artery reactivity will be assessed by ultrasound and FMD will be calculated as the change in brachial artery diameter after release of suprasystolic blood pressure cuff inflation. A blood pressure cuff will be inflated on the upper arm to induce increase in blood flow, termed reactive hyperemia, which increases arterial diameter. The change in vessel diameter is determined by high-resolution ultrasound imaging. The endothelium-dependent FMD of the brachial artery is quantified as the maximum percent change in arterial diameter, expressed in units of "% of brachial artery".
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: % of brachial artery diameter
Arm/Group | Lovaza | Placebo
Number analyzed (Participants) | 39 | 39
% of brachial artery diameter | 6.4 (5.9) | 7.5 (3.1)

ADVERSE EVENTS:
Time Frame: AE reporting lasted the duration of the study (28 weeks)
Groups:
- Lovaza-Active: Lovaza, dietary counseling
Arm/Group | Lovaza-Active | Placebo
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 29/41 | 29/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovaza-Active (N=41) | Placebo (N=41)
loose stool (Gastrointestinal disorders) | 4 (4) | 1 (1)
flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
cold (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
early satiety (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastroenteritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
hiccups (Gastrointestinal disorders) | 1 (1) | 0 (0)
renal stone (Renal and urinary disorders) | 2 (2) | 0 (0)
worsening diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
fish burps (Gastrointestinal disorders) | 2 (2) | 0 (0)
lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
GI blockage (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 1 (1) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
fish taste (Gastrointestinal disorders) | 0 (0) | 2 (2)
anal polyp surgery (Gastrointestinal disorders) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 0 (0) | 1 (1)
heart burn (Gastrointestinal disorders) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
oral thrush (Gastrointestinal disorders) | 0 (0) | 1 (1)
enlarged aorta (Cardiac disorders) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
testosterone insufficiency (Reproductive system and breast disorders) | 0 (0) | 1 (1)
insomnia (Nervous system disorders) | 0 (0) | 1 (1)
nodule under chest (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
nodule right carotid (Cardiac disorders) | 0 (0) | 1 (1)
knee replacement (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
We had low numbers that may not represent the overall population. There was not an HIV negative control arm. The 4 week wash out was too short and therefore difficult to compare the post-treatment vs true post placebo effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less